CLINICAL TRIAL: NCT06736418
Title: A Phase 1a/b, Open-label, Dose-escalation Study of the Safety, Pharmacokinetics, and Initial Efficacy of 225Ac-ABD147 in Patients With Small Cell Lung Cancer and Large Cell Neuroendocrine Carcinoma of the Lung Following Platinum-based Chemotherapy
Brief Title: Study of 225Ac-ABD147 to Establish Optimal Dose in Patients With SCLC and LCNEC of the Lung That Previously Received Platinum-based Chemotherapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abdera Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 225Ac-ABD147-101
Record Dates: First submitted 2024-11-21; First posted 2024-12-16 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Small-Cell Lung Cancer (SCLC); Large Cell Neuroendocrine Carcinoma of the Lung
Keywords: Actinium; Ac-225; 225Ac-ABD147; Indium; In-111; 111In-ABD147; ABD147; Abdera Therapeutics; Abdera; ROVEr; Ac; In; ABD-147; Small Cell Lung Cancer; Small-Cell Lung Cancer; SCLC; Large Cell Neuroendocrine Carcinoma; Large-Cell Neuroendocrine Carcinoma; LCNEC; Lung Cancer; Delta-Like Ligand 3; Delta Like Ligand 3; Delta-Like Protein 3; Delta Like Protein 3; Delta-Like Canonical Notch Ligand 3; Delta Like Canonical Notch Ligand 3; Delta3; DLL3; Precision Radiopharmaceutical; Radiopharmaceutical; Radiotherapy; Radioligand; Linker-Chelator; Linker Chelator; VHH-Fc; HH-FcRN; Biologic; Antibody; Antibodies; Nuclide
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose Escalation and Dose Expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a Dose Escalation Group (Experimental): 225Ac-ABD147 administered in escalating dose cohorts
  Interventions: Drug: 225Ac-ABD147
- Phase 1b Dose Expansion Group (Experimental): Expansion Dose Level selected from Phase 1a Dose Escalation
  Interventions: Drug: 225Ac-ABD147

INTERVENTIONS:
Drug: 225Ac-ABD147 — A delta-like ligand 3 (DLL3)-targeting antibody fragment conjugated with a linker-chelator that effectively coordinates Ac-225

SUMMARY:
The study has 2 parts, Phase 1a and Phase 1b. The goal of Phase 1a is to gather safety, PK and initial efficacy data for 225Ac-ABD147 to better understand best doses for patients with small cell lung cancer (SCLC) and large cell neuroendocrine carcinoma (LCNEC) of the lung following platinum-based chemotherapy.

An initial group of patients will also be given an experimental imaging agent called 111In-ABD147 to help understand where ABD147 goes in the body.

The goal of Phase 1b is to gather additional safety and efficacy data on 225Ac-ABD147 to determine the best dose and to understand how those doses affect the same types of patients' cancers explored enrolled in Phase 1a.

DETAILED DESCRIPTION:
This is an open-label, Phase 1a/b, first-in-human study to assess the safety profile, tolerability, biodistribution, pharmacokinetics (PK), and preliminary antitumor activity of 225Ac-ABD147 in patients with confirmed locally advanced or metastatic small cell lung cancer (SCLC) and large cell neuroendocrine carcinoma (LCNEC) of the lung. All patients must have previously received platinum-based chemotherapy.

Phase 1a will determine the safety, tolerability, dosimetry, PK, and the dose of 225Ac-ABD147 for expansion in the Phase 1b portion.

In addition to receiving treatment, a subset of patients in Phase 1a will undergo either 111In-ABD147-based or 225Ac-ABD147 dosimetry assessments to confirm tumor specificity, identify biodistribution, and to provide insight into dose absorption into tumor and normal tissues.

Phase 1b will evaluate the safety and preliminary efficacy of 225Ac-ABD147 as based on the Phase 1a dose level for expansion by the Safety Review Committee to determine the recommended Phase 2 dose (RP2D).

ELIGIBILITY:
Key Inclusion Criteria:

* Has confirmed, locally advanced or metastatic SCLC or LCNEC of the lung.
* Has completed platinum-based chemotherapy.
* Mentally competent and able to understand and sign an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved Informed Consent Form (ICF)prior to any study specific evaluation.
* Age ≥18 years old at the time the ICF is signed.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 2.
* Expected life expectancy of >12 weeks per the Investigator.
* Has disease that is measurable by RECIST v 1.1.
* Patients with known brain metastases are eligible provided they are considered by the Investigator to be neurologically stable and meet the following criteria: a. Radiotherapy or surgery for brain metastases was completed at least 2 weeks prior to Cycle 1 Day 1 (C1D1); b. Symptoms are stable and steroid/antiepileptic doses remain unchanged for a minimum of 2 weeks prior to C1D1.
* At least 4 weeks from prior major surgery (other than for brain metastases), or at least 7 days from prior non-study-related minor surgery prior to C1D1. In all cases, patient must be sufficiently recovered and stable before study treatment administration.
* Willing to provide archival tumor tissue for central analysis; if unavailable, a pre-study treatment biopsy may be collected and provided.
* Female and male patients of childbearing potential agree to use at least 2 highly effective forms of contraception (1 at least must be barrier method) or agree to completely remain abstinent for duration of study and for 6 months after the last administration of study drug for both female patients and male patients.
* Patients agree to not make semen/egg donations during treatment, within 2 weeks following the last dose of 111In-ABD147, and for 6 months following the last dose of 225Ac-ABD147.

Key Exclusion Criteria:

* Was previously treated with 225Ac-ABD147.
* Has a history of steroid dependent hepatitis caused by treatment with a checkpoint inhibitor.
* Is actively enrolled in another clinical study unless it is an observational (noninterventional) clinical study or the follow-up component of an interventional study.
* Use of an anticancer therapy, radiotherapy (external beam radiotherapy [EBRT], brachytherapy, inoperative radiation therapy, radiopharmaceuticals), or immunotherapy within 3 weeks prior to C1D1. Prior treatment with DLL3-targeting agent is acceptable with appropriate washout.
* Has a medical history of myocardial infarction or unstable angina within 6 months before C1D1.
* Has clinically significant cardiac disease not controlled on medical therapy (eg, congestive cardiac failure, arrhythmia, coronary heart disease).
* Has evidence of active infection requiring intravenous (IV) antibiotics during Screening requiring therapy within 7 days prior to C1D1.
* Has active uncontrolled bleeding or a bleeding diathesis within 28 days prior to C1D1.
* Has serious or non-healing wound, fistula, skin ulcer, or non-healing bone fracture within 7 days prior to C1D1.
* Has received any thoracic radiotherapy within 8 weeks prior to C1D1.
* Has a history of idiopathic pulmonary fibrosis, organizing pneumonia (eg, bronchiolitis obliterans), drug-induced pneumonitis (requiring steroids or immunosuppressive agents), or idiopathic pneumonitis, or evidence of active pneumonitis on the Screening chest computed tomography (CT) scan. Note: History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Has known hypersensitivity to Ac-225; for patients participating in the 111In-ABD147 dosimetry substudy, also has known hypersensitivity to In-111.
* Has known hypersensitivity to Chinese hamster ovary cell products.
* Has a history of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
* Has human immunodeficiency virus infection; patients who are taking an effective antiviral therapy with undetectable viral load prior to C1D1 are eligible.
* Has chronic hepatitis B virus (HBV) infection. Patients who are taking an effective suppressive therapy and have an undetectable HBV viral load are eligible.
* Has a history of hepatitis C virus (HCV) infection, unless treated and cured; patients with HCV infection who are currently on treatment and have an undetectable HCV viral load are eligible.
* Has carcinomatous meningitis.
* Has active symptomatic cord compression.
* Has active symptomatic superior vena cava syndrome.
* Has another primary malignancy that has not been treated with curative intent (discuss with Medical Monitor), except for non-metastatic cutaneous basal cell or squamous cell carcinoma, or non-muscle invasive bladder cancer.
* Is unwilling or unable to follow protocol requirements.
* Has any condition that, in the opinion of the Investigator, would interfere with evaluation of the investigational product or interpretation of the patient's safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Ph 1a: Safety of 225Ac-ABD147 - Number and Grade of Adverse Events | 12 months
  Incidence of adverse events and serious adverse events graded according to NCI-CTCAE v5.0; Clinically significant changes from baseline for laboratory values, ECGs, and vital signs will be evaluated as adverse events.
Ph 1a: Tolerability of 225Ac-ABD147 - Number of Dose Limiting Toxicities | 12 months
  Incidence and nature of dose limiting toxicities.
Ph 1b: Safety of 225Ac-ABD147 to Determine the RP2D for Further Development - Number and Grade of Adverse Events | 12 months
  Incidence of adverse events and serious adverse events graded according to NCI-CTCAE v5.0; Clinically significant changes from baseline for laboratory values, ECGs, and vital signs will be evaluated as adverse events.
Ph 1b: Preliminary Efficacy of 225Ac-ABD147 - Overall Response Rate (ORR) | 12 months
  ORR of confirmed complete response (CR) and partial response (PR) per investigator assessment using RECIST v1.1.
Ph 1b: Preliminary Efficacy of 225Ac-ABD147 - Disease Control Rate (DCR) | 12 months
  DCR per investigator assessment using RECIST v1.1.
Ph 1b: Preliminary Efficacy of 225Ac-ABD147 - Duration of Response (DOR) | 12 months
  DOR of confirmed CR and PR per investigator assessment using RECIST v1.1.
Ph 1b: Preliminary Efficacy of 225Ac-ABD147 - Duration of Progression Free Survival (PFS) | 12 months
  PFS per investigator assessment using RECIST v1.1.
Ph 1b: Preliminary Efficacy of 225Ac-ABD147 - Overall Survival (OS) | 12 months
  OS.
Ph 1b: Preliminary Efficacy of 225Ac-ABD147 - PFS Rate | 12 months
  6 monthly PFS rate per investigator assessment using RECIST v1.1.
Ph 1b: Preliminary Efficacy of 225Ac-ABD147 - OS Rate | 12 months
  6 monthly OS rate.
Ph 1b: Biodistribution and Absorbed Dose - Measurement of Activity | 6 months
  Whole blood radioactivity with whole blood gamma counting.
Ph 1b: Immunogenicity of 225Ac-ABD147 - Measurement of Anti-drug Antibodies | 6 months
  Anti-drug antibody to ABD147.

SECONDARY OUTCOMES:
Ph 1a: Determination of 225Ac-ABD147 Dose for Expansion (Phase 1b) | 12 months
  The dose for expansion (Phase 1b) will be determined by integrating the totality of data obtained in Phase 1a.
Ph 1a: Safety and Tolerability of Multiples Doses of 225Ac-ABD147 - Number and Grade of Adverse Events | 12 months
  Incidence of adverse events and serious adverse events graded according to NCI-CTCAE v5.0; Clinically significant changes from baseline for laboratory values, ECGs, and vital signs will be evaluated as adverse events.
Ph 1a: PK Profile of 225Ac-ABD147 - Peak Plasma Concentration (Cmax) | 6 months
  Cmax.
Ph 1a: PK Profile of 225Ac-ABD147 - Area under the plasma concentration versus time curve (AUC) | 6 months
  AUC.
Ph 1a: PK Profile of 225Ac-ABD147 - Volume of Distribution (Vd) | 6 months
  Vd.
Ph 1a: PK Profile of 225Ac-ABD147 - Elimination | 6 months
  Half-life.
Ph 1a: PK Profile of 225Ac-ABD147 - Elimination | 6 months
  Clearance.
Ph 1a: Immunogenicity of 225Ac-ABD147 - Measurement of Anti-drug antibodies | 6 months
  Anti-drug antibody to ABD147.
Ph 1a: Safety of 111In-ABD147 - Number and Grade of Adverse Events | 2 weeks
  Incidence of adverse events and serious adverse events graded according to NCI-CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Guanying Wang, MD, MS, Study Director — Abdera Therapeutics Inc.
Locations (5):
- United States (5):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - United Theranostics, Glen Burnie, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah